CLINICAL TRIAL: NCT05914181
Title: How Self-disclosure Influences Reproductive Concerns Among Young Male Cancer Patients? The Mediating Role of Perceived Social Support
Brief Title: The Relationship Between Self-disclosure, Perceived Social Support and Reproductive Concerns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 20230614
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Survivors of Young Male Cancer Survivors
Keywords: reproductive concerns; young male cancer survivors; self-disclosure; perceived social support

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants were recruited from oncology units in two hospitals in Shanxi, China using a convenience sampling.Data were collected using a self-report questionnaire consisting of demographic and disease-related characteristics, and instruments measuring self-disclosure, social support and reproductive concerns.

ELIGIBILITY:
Inclusion criteria : ① male; ② Age 18-40 years old; ③ Diagnosed with cancer for 1 year or more; ④ Know the disease; ⑤ Clear mind, able to understand and cooperate with the investigation; ⑥ Sign informed consent to participate in the study voluntarily. Exclusion criteria: ① There were serious primary diseases of liver, kidney, hematopoietic, and serious organ failure; ② He has a history of mental illness, personality disorder, cognitive impairment, and organic brain disease.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants were recruited from oncology units in two hospitals in Shanxi, China using a convenience sampling. The eligible participants were invited to complete the questionnaire after they agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Participants characteristics | once
  Demographic and disease related characteristics included age, marital status, fertility status, payment method of medical expenses, primary caregiver, family history, treatment method, fertility intention, etc.
self-disclosure | once
  Distress Disclosure Index (DDI) was used to evaluated the level of self-disclosure of young male cancer patients
perceived social support | once
  the Perceived Social Support Scale (PSSS) was used to evaluate the level of perceived social support of young male cancer patients which includes 3 dimensions which are named by friend support, family support and other support, with a total of 12 items.
reproductive concerns | once
  the Reproductive concerns after cancer scale-male（RCAC-M） was used to evaluata the level of reproductive concerns in young male cancer survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhao, Study Director — The First Affiliated Hospital of Soochow University
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu L, Chen X, Dong T, Yan W, Wang L, Li W. Self-disclosure, perceived social support, and reproductive concerns among young male cancer patients in China: A mediating model analysis. Asia Pac J Oncol Nurs. 2024 May 4;11(7):100503. doi: 10.1016/j.apjon.2024.100503. eCollection 2024 Jul. PMID 39072257